CLINICAL TRIAL: NCT05529199
Title: Impact of Preoperative Hypocaloric Hyperproteinic Lipid Restricting Diet on Bariatric Surgery
Acronym: LipiDiet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8689
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Obesity, Abdominal
Keywords: Obesity, Abdominal; Preoperative diets; PSMF diet
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity is one of the greatest pandemics of the 21st century with 30 million new cases each year. In France each year, 60,000 bariatric surgery procedures are performed.

Many preoperative diets have been proposed in the literature with some studies giving positive results. But these diets are often strict and can have adverse effects on metabolism. Very few studies have described the PSMF diet. The hypothesis would be that this diet is associated with a reduction in liver volume with a reduction in steatosis.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Man and woman
* Patient operated on at the HUS between 2010 and 2021 for bariatric surgery
* Patient not objecting to the reuse of their data for scientific research purposes.

Exclusion criteria:

- Patient who has expressed his opposition to the reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) operated on at the HUS between 2010 and 2021 for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 776 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
liver volume measurement in cm | Files analysed retrospectively from Ocober 01, 2010 to December 31, 2021 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Benoit ROMAIN, MD, PhD, Principal Investigator — Service de chirurgie générale et digestive - CHU de Strasbourg - France
Locations (1):
- Service de chirurgie générale et digestive - CHU de Strasbourg - France, Strasbourg, France